CLINICAL TRIAL: NCT04904796
Title: Effects of Constraint-induced Movement Therapy With Home-based Hand-arm Bimanual Intensive Therapy in Real-world Bimanual Hand Use in Children With Unilateral Cerebral Palsy
Brief Title: Effects of Constraint-induced Movement Therapy With Home-based Hand-arm Bimanual Intensive Therapy in Children With Unilateral Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeong Yi Kwon, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SMC 2021-04-042
Record Dates: First submitted 2021-05-23; First posted 2021-05-27 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Cerebral Palsy, Spastic Hemiplegic
Keywords: Constraint-Induced Movement Therapy; Home-based Hand-arm Bimanual Intensive Therapy; Unilateral Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Constraint-induced Movement Therapy With Home-based Hand-arm Bimanual Intensive Therapy (Experimental): Children in experimental group will receive 2-hour clinic-based CIMT sessions, 5 days/week for 3 weeks (30 hours), and 2-hour home-based HABIT sessions, 3 days/week for 5 weeks (30 hours).
  Interventions: Other: CIMT; Other: H-HABIT
- Constraint-induced Movement Therapy only (Active Comparator): Children in experimental group will receive 2-hour clinic-based CIMT sessions, 5 days/week for 3 weeks (30 hours).
  Interventions: Other: CIMT

INTERVENTIONS:
Other: CIMT — CIMT : Constraint-Induced Movement Therapy (CIMT) is a deviation from traditional treatments, used to treat hemiplegia. Its aim is to stimulate the functional use of the affected limb and reverse the process developmental is disregard. In this method, the unaffected or less affected limb is restrained, so the person has to use the affected limb.
Other: H-HABIT — H-HABIT : Hand-Arm Bimanual Intensive Therapy (HABIT) in children with hemiplegia is a new intervention developed at Columbia University. HABIT aims to improve the use and coordination of both arms in daily function. Unlike CIMT, HABIT focuses on improving the ability to perform bimanual activities. Participants will be monitored via webcam-based software (i.e. ZOOM) while they performed the activities in their own home.
  Arms: Constraint-induced Movement Therapy With Home-based Hand-arm Bimanual Intensive Therapy

SUMMARY:
This study evaluates the therapeutic effects of constraint-induced movement therapy (CIMT) with home-based hand-arm bimanual intensive therapy (H-HABIT) with unilateral cerebral palsy. Half of the participants will receive CIMT and H-HABIT and others will only receive CIMT.

ELIGIBILITY:
Inclusion Criteria:

* Age 4 to 12 years
* MACS level 1-3
* Diagnosed with unilateral CP due to central nervous system lesions

Exclusion Criteria:

* Severe cognitive dysfunction that rendered them unable to perform simple tasks (e.g., reaching, grasping
* Untreated seizures
* Visual or auditory problems interfering with treatment
* Prior history of musculoskeletal disorders.
* MACS level 4-5

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
Change from Assisting Hand Assessment (AHA) score at 2-month follow-up test | baseline and 2 months
  AHA is a standardized tool for children(18 months-12 years) with unilateral CP. The AHA measures the child's ability to use the affected hand to assist the unaffected hand in a variety of bimanual activities. The 15-20 minute session uses semi-structured play with specific items. A certified AHA assessor views the videorecording to score the child's displayed willingness and ability to use the weaker arm and hand on each of 22 items from 1 (= does not do) to 4 (= effective). The AHA has inter- and intra-rater reliabilities of 0.98 and 0.97 respectively and content validity established during initial development. For data analysis, we generated AHA Logit scores (as recommended in the administration manual) that transform the raw (ordinal) scores into interval level data.

SECONDARY OUTCOMES:
Change from Baseline Pediatric Motor Activity Log (PMAL) score at 2-month follow-up test | baseline and 2 months
  The PMAL was derived from the Motor Activity Log, which is used as an assessment tool in adults who participated CIMT, to measure changes in upper extremity use in real life. This parental assessment tool rates the use of the children's affected upper extremities in daily activities. Twenty-two arm-hand functional tasks that are typical for children aged 7 months to 8 years (e.g., taking off socks or shoes, holding a cup) were assessed and collected as a systemic data. The test has two components: (1) how often (PMAL HO) and (2) how well (PMAL HW). Parents rate PMAL HO on a 6-point scale from 0 (not at all) to 5 (all the time) and PMAL HW from 0 (does not use) to 5 (same as the unaffected arm). This tool has a high test-retest reliability (r=0.94; P<0.01) and a high internal consistency (Cronbach's α=0.88 to 0.95).
Change from Baseline Melbourne Assessment 2 (MA2) score at 2-month follow-up test | baseline and 2 months
  The Melbourne Assessment 2 (MA2) is a specific upper limb assessment focusing on the capacity of one hand. It benchmarks against certain criteria, delving into facets like movement range, accuracy, agility, and flow. The test was videotaped for analysis, and the raw score converted to a percentage of the maximal score.The higher the score, the better the motor function is interpreted. Test-retest results revealed moderate to high intrarater reliability for item totals (mean of 0.83 and 0.79) for each rater and high reliability for test totals (0.98 and 0.97).
Change from Canadian Occupational Performance Measure (COPM) score at 2-month follow-up test | baseline and 2 months
  The COPM was designed as an outcome measure with a semi-structured interview format and structured scoring method to assess a person's level of self-efficacy. It conceptualizes self-efficacy in terms of self-perception of performance and satisfaction with performance. The COPM uses three 10-point rating scales to rate importance, performance and satisfaction. A score value of '1' refers to a low rating (i.e. 'not important at all', not able to do it at all', 'not satisfied at all'). A score value of '10' refers to a high rating (i.e. 'extremely important', 'able to do it extremely well', 'extremely satisfied'). Summing the ratings across problems and dividing by the total number of problems derive separate total performance and satisfaction scores.
Change from Pediatric Evaluation of Disability Inventory Computer Adaptive Test (PEDI-CAT) score at 2-month follow-up test | baseline and 2 months
  The Pediatric Evaluation of Disability Inventory Computer Adaptive Test (PEDI-CAT) was developed to respond to the need for an accurate and efficient functional measure with content for children and youth in multiple functional content areas. The new PEDI-CAT measures function in the three domains of Daily Activities, Mobility and Social/Cognitive for infants, children and youth from birth through 20 years of age. In addition, the PEDI-CAT's Responsibility domain measures the extent to which the caregiver or child takes responsibility for managing complex, multi-step life tasks. The higher the score, the better the functional ability is interpreted.
Change from baseline Use ratio(Accelerometer) at 2-month follow-up test | baseline and 2 months
  Use ratio provides a measurement that lets one compare the frequency of activity between the paretic and nonparetic arms: hours of paretic hand use/hours of nonparetic hand use. A use ratio equal to 1 indicates that the paretic and nonparetic arms are used an equal amount of time throughout the day, and values >1 indicates greater use of the paretic arm. To calculate hours of arm movement, the number of epochs with activity counts >0 will be summed and converted to hours for each arm.
Change from baseline Magnitude ratio(Accelerometer) at 2-month follow-up test | baseline and 2 months
  The magnitude ratio is calculated as a metric to compare the magnitude of acceleration of the arms at each time point: ln(paretic magnitude/nonparetic magnitude). The magnitude will be calculated by taking the vector magnitude of the activity counts for each epoch. The natural log will be used to avoid skewness in the ratio caused by an underestimation of the denominator. The average magnitude will be calculated for each period. A magnitude ratio near 0 indicates similar use of each arm, a negative number indicates more use of the nonparetic arm, and a positive number indicates more use of the paretic arm.
Change from baseline Bilateral magnitude(Accelerometer) at 2-month follow-up test | baseline and 2 months
  The bilateral magnitude is used to compare the overall movement of both arms together as a measure of bilateral arm movement: nonparetic magnitude + paretic magnitude. As with the magnitude ratio, the vector magnitude of the activity counts will be calculated for each epoch. A greater bilateral magnitude indicates greater overall movement of both arms.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Hwang Y, Kwon JY. Identifying the most representative actigraphy variables reflecting standardized hand function assessments for remote monitoring in children with unilateral cerebral palsy. BMC Pediatr. 2024 Apr 25;24(1):273. doi: 10.1186/s12887-024-04724-z. PMID 38664706